CLINICAL TRIAL: NCT05430789
Title: Nurse-led Post-discharge Cessation Support for Smoking Patients Using Mobile-based Intervention: a Randomized Controlled Trial
Brief Title: Post-discharge Cessation for Smoking Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Princess Margaret Hospital, Hong Kong (Other Government); Queen Elizabeth Hospital, Hong Kong (Other); Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SC discharge; HKU Clinical Trials Registry (Registry Identifier: 17614621)
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Smoking Cessation; Post-discharge; Mobile Health
Keywords: Behavioral change techniques; Smoking cessation; Mobile health technology; Nurse-led intervention; Post-discharge; Discharged patients
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 5As brief advice + Self-help ebooklet + Nurse-led mHealth intervention
  Interventions: Behavioral: 5As brief advice; Behavioral: Self-help e-booklet; Behavioral: Nurse-led mHealth intervention
- Control group (Active Comparator): 5As brief advice + Self-help ebooklet + Text messaging
  Interventions: Behavioral: 5As brief advice; Behavioral: Self-help e-booklet; Behavioral: Regular intervention

INTERVENTIONS:
Behavioral: 5As brief advice — Participants will receive brief face-to-face advice following a 5As model at baseline:
  1. Ask: Smoking patients will be asked about their smoking status.
  2. Advise: Smoking patients will be advised to quit in a clear and personalised manner, with a focus on smoking-related diseases.
  3. Assess: Smoking patients will be assessed for their readiness to quit by assessing their self-efficacy and perceived importance.
  4. Assist: Those who are ready to quit will be assisted in setting a quit plan.
  5. Arrange: Refer to smoking cessation services.
Behavioral: Self-help e-booklet — A 12-page generic self-help smoking cessation e-booklet via IM apps, including:
  1. Highlights of the absolute risk of death due to smoking;
  2. Smoking and diseases management;
  3. Ten horrible pictorial warnings of health consequences of smoking and second-hand smoking;
  4. Benefits of quitting;
  5. Methods to quit and handle. withdrawal symptoms.
Behavioral: Nurse-led mHealth intervention — Participants will receive real-time mHealth behaviour and psychosocial support for 12 weeks after baseline through IM apps. mHealth intervention consists of two main parts: regular instant messaging on smoking cessation and personalized real-time mHealth chatting on smoking and disease (including active referral to smoking cessation service)
  Arms: Intervention group
Behavioral: Regular intervention — Participants will receive text messages using IM app with content on general health and reminding the importance of participating in the follow-up surveys and biochemical validation for quitting.
  Arms: Control group

SUMMARY:
This study aims to enhance the general 5As brief advice model with interactive mobile phone-based intervention and active referral to community smoking cessation services for smoking patients discharged from hospitals.

DETAILED DESCRIPTION:
Most smoking patients continue to smoke (76.1%) after being discharged from hospitals. Post-discharge smoking cessation (SC) support is one of the most cost-effective treatments. Hospitalisation offers a teachable moment to motivate patients to engage in post-discharge intervention, particularly those suffering from smoking-related diseases. Behavioral and psychosocial support increases abstinence in patients. Current clinical guidelines in the US (USPSTF) and UK (NICE) recommend health care professionals to provide brief SC support to patients using a brief advice model such as the 5As (Ask, Assess, Advice, Assist, Arrange) and further motivational 5Rs interventions (Relevance, Risks, Rewards, Roadblocks, and Repetition) if needed for those not having quit attempts. A key trial found that providing discharged patients with such proactive and sustained care as free SC medication, telephone calls to promote quitting, and additional counselling through clinic referrals increased 6-months validated quitting. Trained patient navigators providing patients in hospital primary clinics with tailored individual advice with medication and counselling referrals were found to be effective at improving 12-months quitting. Previous trials also showed connecting community smokers or smokers who visited emergency departments to existing SC services increased validated quitting at 6-months. Recent advances in mobile phone technology allow incorporating such innovations to improve the cost-effectiveness of post-discharge smoking cessation services.

Mobile phones are increasingly used for monitoring and delivering personalised health treatments (mHealth). Regular text messaging was found to increased 6-months validated abstinence in general smokers, although the study was limited to pre-defined messages and interactions. A previous study reported an automated interactive voice response to be favored by patients and to increase abstinence. A text-based programme was tested in a Chinese population, and previous study found the delivery of interactive chat-based SC support via IM apps to be effective in increasing quitting. Chat-based SC interventions can provide real-time, personalised behavioral support and referrals to SC services. Mobile health is also part of the World Health Organization's strategies to combat smoking.

Leveraging the success of previous trials in inpatients and a chat-based trial using IM to deliver behavioral support to community smokers, This study proposes to refine the 5As cessation model by incorporating a mobile phone-based intervention for patients recently discharged from hospitals. Recent trials showed a mobile phone-delivered cessation intervention combined with SC medication service increased abstinence. Recent trials showed a mobile phone-delivered cessation intervention combined with SC medication service increased abstinence. Active referral of community smokers to smoking cessation services increases service use and quitting but smoking patients were not referred for sustained cessation service in hospitals in Hong Kong. The effect of mobile phone-based intervention with active referral to link discharged patients for standard smoking cessation service remains unclear. Therefore, This study proposes to enhance the general 5As brief advice model with interactive mobile phone-based intervention and active referral to community smoking cessation services for smoking patients discharged from hospitals in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

1. Smokers who are hospitalised or waiting for discharge in Hong Kong
2. Smoke cigarettes or alternative tobacco products (e.g. electronic cigarettes or heated tobacco products) daily at 1 month prior to hospitalisation
3. Have a smartphone with an IM app (WhatsApp or WeChat) and experience in using the app
4. Hong Kong adult residents (18+) able to communicate in Chinese (Cantonese or Mandarin)

Exclusion Criteria:

1. Smokers not mentally fit for communication (e.g. psychiatry patients)
2. Smokers currently using SC medication or other SC services
3. Smokers hospitalised for more than 1 month
4. Perceived difficulty to use IM after discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Biochemically-validated abstinence | 6-month after baseline
  Defined by exhaled carbon monoxide < 4 parts per million (ppm) and salivary cotinine < 30 ng/ml
Biochemically-validated abstinence | 12-month after baseline
  Defined by exhaled carbon monoxide < 4 parts per million (ppm) and salivary cotinine < 30 ng/ml

SECONDARY OUTCOMES:
Self-reported past 7-day abstinence | 6-month after baseline
  Being completely smoke-free in the past 7 days
Self-reported past 7-day abstinence | 12-month after baseline
  Being completely smoke-free in the past 7 days
24-weeks continuous abstinence | 6-month after baseline
  Being completely smoke-free in the past 24 weeks
24-weeks continuous abstinence | 12-month after baseline
  Being completely smoke-free in the past 24 weeks
Intention to quit | 6-month after baseline
  A single item will measure if smokers plan to quit smoking in 30 days, with response of yes or no
Intention to quit | 12-month after baseline
  A single item will measure if smokers plan to quit smoking in 30 days, with response of yes or no
Number of quit attempt | 6-month after baseline
  Defined by abstinence for at least 24 hours
Number of quit attempt | 12-month after baseline
  Defined by abstinence for at least 24 hours
Smoking reduction | 6-month after baseline
  Defined by at least 50% self-reported reduction in baseline daily number of cigarettes
Smoking reduction | 12-month after baseline
  Defined by at least 50% self-reported reduction in baseline daily number of cigarettes
Nicotine dependence level | 6-month after baseline
  Assessed by Heaviness of Smoking Index (range 0 to 6 with higher score indicating greater nicotine dependence)
Nicotine dependence level | 12-month after baseline
  Assessed by Heaviness of Smoking Index (range 0 to 6 with higher score indicating greater nicotine dependence)
Smoking cessation service use | 6-month after baseline
  Any access to a smoking cessation service
Smoking cessation service use | 12-month after baseline
  Any access to a smoking cessation service

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No